CLINICAL TRIAL: NCT07293325
Title: Assessing the Role of GLP-1 Receptor Agonist Semaglutide and Dual GLP-I/GIP Receptor Agonist Tirzepatide in Delaying Genetic Aging in Adult Obese Patients Using the iWatchAge Technology
Brief Title: Semaglutide and Tirzepatide for Genetic Aging Delay in Adults With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0568
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-06

CONDITIONS: Adults With Simple Obesity
MeSH Terms: interventions — semaglutide; Tirzepatide; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Semaglutide Group (Experimental): Semaglutide administered once weekly by subcutaneous iniection. Dose titrated from 0.25 mg to 2.0 mg as tolerated over 24 weeks
  Interventions: Drug: Semaglutide
- Tirzepatide Group (Experimental): Tirzepatide administered once weekly by subcutaneous injection. Dose titrated from 2.5 mg to 10 mg as tolerated over 24 weeks
  Interventions: Drug: Tirzepatide
- Metformin Group (Active Comparator): Metformin administered orally. Dose titrated from 500 mg to 1500-2000 mg daily, based on tolerance, for 24 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Semaglutide — Semaglutide administered once weekly by subcutaneous injection.Dose titrated from 0.25 mg to 2.0 mg as tolerated over 24 weeks
  Arms: Semaglutide Group
Drug: Tirzepatide — Tirzepatide administered once weekly by subcutaneous injection. Dose titrated from 2.5 mg to 10 mg as tolerated over 24 weeks
  Arms: Tirzepatide Group
Drug: Metformin — Metformin administered orally. Dose titrated from 500 mg to 1500-2000 mg daily, based on tolerance, for 24 weeks
  Arms: Metformin Group

SUMMARY:
This study is a prospective, randomized, open-label clinical trial enrolling 66 adults with simple obesity who have not used weight-loss medications for at least 3 months. Participants will receive semaglutide, tirzepatide, or metformin for 24 weeks. Changes in "biological (epigenetic) age" will be assessed using the iWatchAge DNA methylation age test, while simultaneously monitoring improvements in aging-related biomarkers such as inflammatory factors, metabolic parameters, and body composition. The aim is to determine whether incretin-based therapies can reverse or slow obesity-related accelerated epigenetic aging and to provide new clinical evidence for interventions targeting obesity and aging.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 75 years.
2. Diagnosed with simple obesity, defined as BMI ≥ 30 kg/m².
3. Have not used any anti-obesity medications (including GLP-1 RAs, tirzepatide, metformin for weight loss, etc.) within the past 3 months.
4. Able and willing to comply with study procedures and complete follow-up assessments.
5. Provide written informed consent.

Exclusion Criteria:

1. Presence of secondary obesity (e.g., endocrine disorders such as Cushing's syndrome or hypothyroidism).
2. Use of anti-obesity medications or participation in another weight-loss program within the past 3 months.
3. Diagnosed type 1 or type 2 diabetes mellitus requiring hypoglycemic drug therapy.
4. History of pancreatitis, severe gastrointestinal disease, or bariatric surgery.
5. Severe cardiovascular, hepatic, renal, or psychiatric disease that may affect participation.
6. Pregnant or breastfeeding women, or women planning pregnancy during the study period.
7. Current participation in any other clinical trial.
8. Any condition that, in the investigator's judgment, makes the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-04-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Change in DNA methylation-based biological age measured by iWatchAge | Baseline and Week 24
  Change in epigenetic biological age from baseline to Week 24, measured using the iWatchAge DNA methylation assay. This outcome reflects whether semaglutide, tirzepatide, or metformin can delay or reverse obesity-associated accelerated epigenetic aging.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China